CLINICAL TRIAL: NCT04156204
Title: Kidney Immunosuppression Dosed Daily Only (KIDDO) - A Pilot Study
Brief Title: Immunosuppressant Medication Dosed Daily After Kidney Transplant
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Discontinuation of study due to site staffing and resources available to conduct the study
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-2311
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Kidney Transplant Rejection; Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Longitudinal Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adolescent and Young Adult (AYA) Kidney Transplant Recipients (Experimental): AYA kidney transplant recipients will receive a Medication Event Monitoring System (MEMS) in the form of a medication bottle and cap system and once daily tacrolimus XR 1-10mg
  Interventions: Other: Medication Event Monitoring System (MEMS); Drug: Once-Daily Tacrolimus extended release

INTERVENTIONS:
Other: Medication Event Monitoring System (MEMS) — AYA kidney recipients will receive a Medication Event Monitoring System (MEMS) via medication bottle and cap system
Drug: Once-Daily Tacrolimus extended release — AYA kidney recipients will receive once daily tacrolimus XR 1-10mg daily
  Other Names: Envarus XR

SUMMARY:
Medication non-adherence is a major risk factor for graft dysfunction and graft loss among pediatric and adult transplant recipients. Rates of non-adherence in these populations are estimated between 30 and 70%, with the highest prevalence in adolescent and young adult (AYA) transplant recipients. Treatment-related factors known to impact rates of adherence include the number of medication doses per day and the number of tablets or capsules a patient takes per day, or "pill burden". One approach to minimizing dosing frequency and pill-burden includes transitioning patients to once-daily formulations. The current literature investigating utilization of once-daily immunosuppressive regimens in the AYA kidney transplant population is limited.

DETAILED DESCRIPTION:
One approach to minimizing dosing frequency and pill-burden includes transitioning patients to once-daily formulations.3 The current literature investigating utilization of once-daily immunosuppressive regimens in the AYA kidney transplant population is limited. Two studies have demonstrated safe and effective conversion of twice-daily tacrolimus to the Astagraf® in stable pediatric solid organ transplant recipients.4,5 Patients maintained equivalent tacrolimus exposure and experienced similar rates of rejection and graft loss in the first year post-conversion.5 To date, experience with another once-daily extended release (XR) tacrolimus product, Envarsus XR®, has not been published in the AYA population. Additionally, adherence studies evaluating a once-daily immunosuppression regimen including extended-release tacrolimus and azathioprine (which is dosed once daily as opposed to the twice daily dosing required for azathioprine's alternative mycophenolate mofetil) have not been conducted.

Of note, and even though twice-daily mycophenolate has been shown to be superior to once-daily azathioprine early post-transplant, more long-term data suggest that this advantage may not persist.6 Furthermore, a recent Cochrane review addressed the question of mycophenolate versus azathioprine as primary anti-proliferative immunosuppression for kidney transplant recipients; it concluded that "balancing the benefits and harms of the two drugs remains a major task of the transplant physician to decide which agent" is appropriate for the individual patient. 7 Moreover, once-daily immunosuppression with tacrolimus extended-release and once-daily azathioprine has been used with excellent results at a British center that focusses on AYA kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-22 years
2. Tanner stage 4/5
3. "Stable" kidney transplant status, as determined by the primary transplant team
4. At minimum 1 year post-kidney transplant or patients meeting all of the above inclusion criteria except 4) who have instead been transitioned to azathioprine by the primary transplant team due to intolerability of mycophenolate mofetil secondary to adverse medication effects (i.e. neutropenia, gastrointestinal intolerance etc.)

Exclusion Criteria:

1. < Tanner stage 4
2. Kidney transplant performed at an institution other than Children's Hospital Colorado, Lurie Children's Hospital of Chicago, or Cincinnati Children's Hospital
3. Recipients of dual solid organ transplants (i.e. heart kidney, liver kidney).

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life: as assessed by change in PedsQL | Day 0, Day 60, Day 210
  Pediatric Quality of Life (PedsQL) Transplant Module Version 3.0 will be used to assess quality of life prior to and after transition from twice to once daily immunosuppressant medication regimen. Health-related quality of life (HRQOL) has been defined as an individual's subjective experience of their illness, and the impact that illness and its treatment have on the individual's functioning in a variety of domains. The PedsQL is a 46-item self- and parent-report measure that rates HRQOL in 8 domains (medication adherence, medication side-effects, social relationship, physical discomfort, worries regarding health status, treatment anxiety, impact on appearance, and communication). The PedsQL Transplant Module assesses physical functioning, emotional functioning, social functioning, and school functioning and was developed through focus groups, cognitive interviews, pretesting, and field testing measurement development protocols. Higher scores indicate lower problems.
Adherence to medical therapies and medications: as assessed by Medication Event Monitoring System (MEMS) at Day 30 | Day 30
  MEMS data will be accessed prior to transition to once-daily medications (baseline adherence) and analyzed accordingly. Dates and times in which medication bottles were opened will be recorded.
Adherence to medical therapies and medications: as assessed by Medication Event Monitoring System (MEMS) at Day 60 | Day 60
  MEMS data will be accessed the first month of transition to once-daily medications (intervention adherence) and analyzed accordingly. Dates and times in which medication bottles were opened will be recorded.
Adherence to medical therapies and medications: as assessed by Medication Event Monitoring System (MEMS) at Day 210 | Day 210
  MEMS data will be accessed 6 months after transition to once-daily medications (retention adherence) and analyzed accordingly. Dates and times in which medication bottles were opened will be recorded.
Adherence to medical therapies and medications: as assessed by Change in Tacrolimus Trough Concentration Variance | Day 0, Day 30, Day 60, and Day 240
  Tacrolimus trough goals between 4-7ng/mL as per Transplant Immunosuppression Protocols. Student T-test, repeated measures for parametric data).
  The standard deviation of tacrolimus troughs will be calculated from the 4 tacrolimus trough values obtained for clinical care purposes preceding Study Visit 1 (SD1). The standard deviation of tacrolimus troughs will be calculated again from the 4 tacrolimus trough values obtained for clinical care purposes preceding Study Visit 4 (SD2).
Adherence to medical therapies and medications:as assessed by Change in Adolescent Medication Barriers Scale (AMBS) | Day 0, Day 60, Day 210
  17 item scale that corresponds to the Parent Medication Barriers Scale (PMBS) with 16 items. Both have strong internal consistency and are scored on a 5-point Likert scale from Strongly Disagree to Strongly Agree. A total score can be calculated, and there are subdomains of disease frustration/adolescent issues, regimen adaptation/cognitive issues, and ingestion issues, with an additional parent reminder domain on the PMBS. Lower scores indicate less barriers to medication adherence.
Adherence to medical therapies and medications: as assessed by Change in The Medical Adherence Measure (MAM) | Day 0, Day 60, Day 210
  Semi-structured interview that has four general modules to assess adherence with medication, diet, exercise, and clinic attendance, as well as illness-specific modules. For the purpose of this study, the Medication and Clinic Attendance Modules will be completed. Non-adherence scores can be calculated based on the degree of adherence on a spectrum of 0%-100% adherent to capture the fluctuations and intricacies of occasional or slightly inconsistent adherence. Missed adherence score = number of doses missed out of the doses prescribed × 100%. Late adherence score = number of doses taken late out of the doses prescribed × 100%, where late is defined as greater than one hour later than the usual routine. Adherence is assessed for each medication separately and then averaged across medications.

SECONDARY OUTCOMES:
Long-term measures of graft and patient survival: as assessed by change in serum creatinine and urinary protein | Day 0, Day 30, Day 60, Day 210, and Day 240
  Markers of graft function will be assessed by measuring levels of serum creatinine and urinary protein. Lower serum creatinine and urinary protein indicate better long-term graft and patient survival.
Long-term measures of graft and patient survival: as assessed by change in markers of proteinuria | Day 30 and Day 210
  Markers of proteinuria will be assessed by urinalysis and random urinary protein/creatinine ratio. Lower urinary protein/creatinine ratio indicates better long-term measures of graft and patient survival.
Long-term measures of graft and patient survival: as assessed by number of episodes of rejection | Up to Day 240
  Graft rejection episodes will be determined to have occurred if indicated by transplant biopsy results. Occurrences of graft rejection episodes among participants will be assessed up to Day 240.
Long-term measures of graft and patient survival: as assessed by change in presence of donor-specific antibody monitoring | Day 0 and Day 240
  Presence of donor-specific antibodies (DSA) prior to and after initiation of intervention.
Long-term measures of graft and patient survival: as assessed by change in presence of BK virus screening results | Day 0 and Day 240
  Includes assessing the viral load to monitor presence of BK virus.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Goebel, MD, Principal Investigator — Children's Hospital Colorado; Mary Chandran, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster BJ, Dahhou M, Zhang X, Platt RW, Samuel SM, Hanley JA. Association between age and graft failure rates in young kidney transplant recipients. Transplantation. 2011 Dec 15;92(11):1237-43. doi: 10.1097/TP.0b013e31823411d7. PMID 22124283
- [Background] Sabaté, E (2003) Adherence to long-term therapies: evidence for action. World Health Organization, Geneva
- [Background] Steinberg EA, Moss M, Buchanan CL, Goebel J. Adherence in pediatric kidney transplant recipients: solutions for the system. Pediatr Nephrol. 2018 Mar;33(3):361-372. doi: 10.1007/s00467-017-3637-0. Epub 2017 Mar 27. PMID 28349215
- [Background] Min SI, Ha J, Kang HG, Ahn S, Park T, Park DD, Kim SM, Hong HJ, Min SK, Ha IS, Kim SJ. Conversion of twice-daily tacrolimus to once-daily tacrolimus formulation in stable pediatric kidney transplant recipients: pharmacokinetics and efficacy. Am J Transplant. 2013 Aug;13(8):2191-7. doi: 10.1111/ajt.12274. Epub 2013 Jun 4. PMID 23734831
- [Background] Heffron TG, Pescovitz MD, Florman S, Kalayoglu M, Emre S, Smallwood G, Wisemandle K, Anania C, Dhadda S, Sawamoto T, Keirns J, Fitzsimmons W, First MR. Once-daily tacrolimus extended-release formulation: 1-year post-conversion in stable pediatric liver transplant recipients. Am J Transplant. 2007 Jun;7(6):1609-15. doi: 10.1111/j.1600-6143.2007.01803.x. PMID 17511684
- [Background] Clayton PA, McDonald SP, Chapman JR, Chadban SJ. Mycophenolate versus azathioprine for kidney transplantation: a 15-year follow-up of a randomized trial. Transplantation. 2012 Jul 27;94(2):152-8. doi: 10.1097/TP.0b013e31825475a3. PMID 22728292
- [Background] Wagner M, Earley AK, Webster AC, Schmid CH, Balk EM, Uhlig K. Mycophenolic acid versus azathioprine as primary immunosuppression for kidney transplant recipients. Cochrane Database Syst Rev. 2015 Dec 3;2015(12):CD007746. doi: 10.1002/14651858.CD007746.pub2. PMID 26633102